CLINICAL TRIAL: NCT06745583
Title: An Open-label, Exploratory, Phase II, Proof-of Concept, Clinical Study to Assess the Safety and Tolerability of EI-1071 in Patients With Alzheimer's Disease (AD)
Brief Title: A Phase 2 Study to Assess the Safety of EI-1071 and the Effects of EI-1071 on Neuroinflammation in Alzheimer's Disease Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Elixiron Immunotherapeutics (Hong Kong) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EI-1071-202; PTC-22-973334 (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Mild, Moderate, or Severe Alzheimer's Disease
Keywords: Alzheimer's Disease; Neuroinflammation; Neurodegenerative Disorder; Cognitive Dysfunction
MeSH Terms: conditions — Lymphoma, Follicular; Alzheimer Disease; Neuroinflammatory Diseases; Neurodegenerative Diseases; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EI-1071 dose (Experimental)
  Interventions: Drug: EI-1071 tablet, oral

INTERVENTIONS:
Drug: EI-1071 tablet, oral — Dose: 448.2 mg BID for 28 days

SUMMARY:
An open-label, exploratory, phase II, proof-of concept, clinical study to assess the safety and tolerability of EI-1071 and the effects of EI-1071 on neuroinflammation in patients with mild, moderate, or severe Alzheimer's disease

DETAILED DESCRIPTION:
This is an open-label, phase II, exploratory, proof-of-concept study to assess the safety and tolerability of EI-1071 and the effects of EI-1071 on neuroinflammation in patients with mild, moderate, or sever Alzheimer's disease (AD). The main goals include:

1. to validate mechanism-engagement of EI-1071 by tracing the change of activated microglia in selected brain regions in AD patients using TSPO PET/MRI imaging.
2. to assess effects of EI-1071 on changes of inflammatory biomarkers associated with AD progression.

ELIGIBILITY:
Inclusion Criteria:

1. Must meet all the clinical criteria for mild to severe AD (i.e., probable or possible AD dementia by NIA-AA criteria; must have objective evidence of cognitive impairment at Screening
2. Clinical Dementia Rating Scale (CDR)≧0.5
3. If using drugs to treat symptoms related to AD, doses must be stable for at least 8 weeks prior to screening.
4. Adequate hematologic, hepatic, and renal function at the screening visit defined by the following criteria:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L
   * Hemoglobin [Hgb] > 10 g/dL
   * Platelet count ≥ 100 × 10⁹/L
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1 × upper limit of normal (ULN)
   * Total bilirubin and direct bilirubin ≤ 1.0 × ULN
   * Alkaline phosphatase (ALP) ≤ 1.0 × ULN
   * Creatinine clearance (CCr) ≥ 60 mL/min
5. Female subject with childbearing potential must have a negative serum pregnancy test at the screening visit (female subjects must be surgically confirmed sterile, i.e., had hysterectomy, bilateral oophorectomy, or tubal ligation procedures), post-menopausal for at least 1 year (documented in the medical history), or must commit to use two contraceptive methods during the study.
6. Female subject with childbearing potential must be willing to implement adequate, highly effective contraceptive measure during the study period. Effective birth control includes:

   * Intrauterine device plus one barrier method
   * Oral, implantable, or injectable contraceptives plus one barrier method; or
   * Two barrier methods

     * Effective barrier methods are male or female condoms, diaphragms, or spermicides (creams or gels that contain a chemical to kill sperm). Women of childbearing potential are those who have not been surgically sterilized or have not been free from menses for ≥ 1 year.
7. Male subject who agrees to use an adequate method of contraception during the study period [e.g., barrier contraceptives (male condom)].
8. Subjects or his/her legal representative or guardian are willing to sign written informed consent and willing to comply with study requirements.

Exclusion Criteria:

1. Body weight ≥ 150 kg or body mass index (BMI) ≥ 35 kg/m² at the screening visit.
2. Prior use of pexidartinib (Turalio), other chemical entities, or any biologic treatment targeting colony stimulating factor 1 (CSF-1) or the CSF-1 receptor within 3-month of the first dose with EI-1071; previous uses of oral tyrosine kinase inhibitors are allowed (e.g., imatinib or nilotinib).
3. AD patients with low binding affinity for tracer TSPO rs6971 SNP polymorphism at screening
4. Pregnant, breast feeding or plan to be pregnant women during the study period
5. Active tuberculosis (TB), active or chronic infection with hepatitis B virus (HBV) or hepatitis C virus (HCV) or known active or chronic infection with human immunodeficiency virus (HIV) at screening or in the medical history.
6. Any medical or neurological/neurodegenerative condition (including mental deficit, intracranial tumor, glioma or meningioma; head trauma, Lewy body dementia; other disease than AD) that, in the opinion of the Investigator, might be a contributing cause to the participant's cognitive impairment or could lead to discontinuation, lack of compliance, interference with study assessments, or safety concerns
7. Clinically significant, unstable psychiatric illness or have contraindications to brain magnetic resonance imaging (MRI) or PET scans
8. Have had a stroke or Transient Ischemic Attack (TIA), unexplained loss of consciousness or relevant brain hemorrhage, bleeding disorder and cerebrovascular abnormalities in the past year based on medical history (with MRI imaging results as confirmation in the medical history) at screening. Subjects with clinically relevant cerebrovascular abnormalities in MRI will be excluded per PI's discretion.
9. Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine (including poor-controlled T2DM), neurological, immunodeficiency, pulmonary, or other disorder or disease at the screening visit (such as neurological or cognitive impairment/decline due to substance abuse, vitamin B12 deficiency, abnormal thyroid function, or other underlying condition might contribute to cognitive, functional or behavioral impairment will be excluded) by investigator's judgment at screening; subjects who have to be fed by enteral tube will be excluded.
10. History of or ongoing malignancy or carcinoma (either concurrent or within the last year of starting study treatment) that requires therapy (e.g., surgical, chemotherapy, or radiation therapy), except for adequately treated basal or squamous cell carcinoma of the skin, melanoma in-situ, carcinoma in-situ of the cervix or breast
11. Currently participating in any other clinical study or have participated in clinical trial within the last 60 days prior to screening; had donated blood (≥ 250 mL) within 30 days at screening.
12. Known allergy to EI-1071 or hypersensitivity to any component of the formulation (e.g., hydroxypropyl methylcellulose acetate succinate) or hypersensitivity to any radiochemical tracer or [¹⁸F]FEPPA radiochemical tracer
13. Required to use strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) and is anticipated to use these inhibitors or inducers during the study period

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 4 [¹⁸F] FEPPA Binding in Selected Brain Regions of Interest | Baseline, Week 4
  Change from baseline in volume of distribution (Vt) of [¹⁸F]FEPPA binding in selected brain regions of interest in each [¹⁸F]FEPPA Positron Emission Tomography (PET) scan obtained from individual patient after 28 days of EI-1071 repeated dosing

SECONDARY OUTCOMES:
Number of Participants With at Least One Adverse Events (AEs) or Serious Adverse Events (SAEs) by CTCAE v5.0 | From Day 1 up to Day 84
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Change From Baseline to Week 12 as Measured by CDR-SB | Baseline, Week 4, Week 12
  CDR was derived through semi-structured interview with the participant and an appropriate informant, and it rated impairment across six domains: memory, orientation, judgment, and problem solving, community affairs, home and hobbies, and personal care on a 5-point scale for which 0=no impairment, 0.5=questionable impairment, and 1, 2, and 3=mild, moderate, and severe impairment, respectively. The CDR-SB is based on
Mean Change From Baseline to Week 12 in Mini Mental State Exam (MMSE) Score | Baseline, Week 4, Week 12
  MMSE is a rater-administered performance-based outcome (PerfO) that includes a set of standardized questions used to evaluate possible cognitive impairment and help stage the severity level of this impairment. The questions target six areas: orientation, registration, attention, short-term recall, language, and constructional praxis/visuospatial abilities. Total score ranges from 0-30, with lower scores indicating greater impairment. A positive change from baseline indicates improvement.
Change From Baseline to Week 12 in Alzheimer Disease Assessment Scale-Cognition Subscale 11 (ADAS-Cog11) Score | Baseline, Week 4, Week 12
  The ADAS-Cog11 was designed to measure cognitive symptom change in participants with Alzheimer's Disease (AD) and consisted of 11 tasks. The standard 11 items (and corresponding score range) were: word recall (0-10), commands (0-5), constructional praxis (0-5), naming objects and fingers (0-5), ideational praxis (0-5), orientation (0-8), word recognition (0-12), spoken language ability (0-5), comprehension of spoken language (0-5), word-finding difficulty (0-5), and remembering test instructions (0-5). The test included 7 performance items and 4 clinician-rated items. The ADAS-Cog11 total score was the sum of all 11 individual items, with a total score ranging from 0 (no impairment) to 70 (severe impairment). Higher scores indicated more severe cognitive impairment. A negative change from baseline indicates improvement.
Change From Baseline to Week 12 in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Total Score | Baseline, Week 4, Week 12
  ADCS-ADL is a 23-item rater-administered, observer-reported outcome (ObsRO) that captures a participant's ability to perform basic activities of daily living (e.g., eating and toileting) and more complex ADL or instrumental activities of daily living (iADL, e.g., using the telephone, managing finances, preparing a meal). Total score ranges from 0-78, with higher scores reflecting better functioning. A positive change from baseline indicates improvement.
Change From Baseline to Week 12 on Behavior in Neuropsychiatric Inventory Questionnaire (NPI-Q) Total Score | Baseline, Week 4, Week 12
  The NPI-Q evaluates 12 neuropsychiatric disturbances common in dementia: delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavioral disturbances and appetite/eating abnormalities. The severity of each neuropsychiatric symptom is rated on a 3-point scale (mild, moderate and marked). The total severity score range is from 0 to 36 with higher scores representing higher severity.
EI-1071 concentrations in plasma | Predose and 2-3 hours post dose in Day1 and Day 14, predose and 2-4 hours post dose in Day 28
  EI-1071 concentrations in plasma samples will be assessed.
EI-1071 concentrations in cerebrospinal fluid | Predose in Day 1 and 2-4 hours post dosing in Week 4
  EI-1071 concentrations in cerebrospinal fluid samples will be assessed.
Neuroinflammation and/or neurodegeneration biomarkers levels in plasma and in cerebrospinal fluid | Predose in Day 1 and 2-4 hours post dose in Day 28
  Neuroinflammation and/or neurodegeneration biomarkers levels in plasma or in cerebrospinal fluid will be assessed.
Physical Examination (PE) | Baseline, Day 1, Week 2, Week 4, Week 8, Week 12
  Clinically significant abnormal changes in physical examinations
Vital Sign | Baseline, Day 1, week 2, week 4, week 8, week 12
  Clinically significant abnormal changes in vital signs
Electrocardiograms (ECGs) changes from baseline for PR | Baseline, Day 1, week 2, week 4, week 8, week 12
  Clinically significant abnormal changes from baseline in ECG for PR
Electrocardiograms (ECGs) changes from baseline for QRS duration | Baseline, Day 1, week 2, week 4, week 8, week 12
  Clinically significant abnormal changes from baseline in ECGs for QRS duration
Electrocardiograms (ECGs) changes from baseline in T wave | Baseline, Day 1, week 2, week 4, week 8, week 12
  Clinically significant abnormal changes from baseline in ECGs in T wave
Electrocardiograms (ECGs) changes from baseline in QTc | Baseline, Day 1, week 2, week 4, week 8, week 12
  Clinically significant abnormal changes from baseline in ECGs in corrected QT interval (QTc)

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No